CLINICAL TRIAL: NCT06156657
Title: Postoperative Efficacy of Subcostal TAP Block in Laparoscopic Sleeve Gastrectomy Surgery: a Randomized Controlled Trial
Brief Title: Postoperative Analgesia of TAP Block for Laparoscopic Sleeve Gastrectomy
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ismail Mohamed Abdelgawad Ahmed, DOCTOR, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAP block
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain
Keywords: subcostal TAP; laparoscopic; sleeve gastrectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anasthesiologist who perform postoperative pain will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP group (Active Comparator): patients candidate for laparoscopic sleeve gastrectomy to receive GA and subcostal TAP block to control postoperative pain and minimize opioid consumption
  Interventions: Other: subcostal TAP block
- Control group (No Intervention): healthy controls candidate for laparoscopic sleeve gastrectomy to receive GA only opioids were used

INTERVENTIONS:
Other: subcostal TAP block — Comparison between subcostal TAP block and opioids for postoperative pain after laparscopic sleeve gastrectomy
  Arms: TAP group

SUMMARY:
many methods were considered to control postoperative pain in laparoscopic bariatic surgery including non steroidal anti-inflammatory drugs, opioids and neuraxial block

but subcostal (TAP) block has provided good analgesic effect when used as a part of multimodal analgesia in bariatric surgery due to lack of visceral block

DETAILED DESCRIPTION:
Since long time opioid have been used to control postoperative pain in bariatric surgery However, an increasing awareness of opioid-related adverse events, including respiratory depression, paralytic ileums, and sedation, constipation has led to a shift towards utilizing opioid-sparing techniques for postoperative analgesia As neuroaxial block and ultrasound guided nerve blocks

As the transverse abdominis plane (TAP) block which is of increasing interest nowadays (Basaran B, et al 2015)

The ultrasound-guided oblique SCTAP block, first described by Hebbard et al., has the potential to provide analgesia for both upper and lower abdominal surgery. There is a growing consensus that the SCTAP block provides better analgesia for upper abdominal incisions

The TAP block via various approaches provides some advantages over neuraxial anesthesia (Ganapathy Set al 2015). For example, TAP blocks are associated with a lower use of intraoperative phenylephrine and a lesser degree of intraoperative blood pressure changes. The SCTAP block may be utilized in cases in which neuraxial anesthesia is contraindicated, such as patients with coagulation issues or infection at the epidural puncture site. Although the SCTAP block provides sensory blockade of the abdominal wall, it is lacking in coverage of visceral pain (Lissauer J,et al 2014).

The lack of visceral pain analgesia may require the use of additional methods of postoperative pain control such as intravenous opioids or non-narcotic analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* ASA Ι-ΙΙ
* BMI >35

Exclusion Criteria:

* Patient refusal.
* Allergy to study drugs.
* Infection at site of injection.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control | 9 months
  by using VAS score

SECONDARY OUTCOMES:
postoperative 24 hour opioid consumption | 9 months
  collecting total doses of opioids consumed in the first 24 hours postoperative in cmparison to the other group
postoperative nausea and vomiting | 9 months
  recording incidence, frequency and severity

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are planned to be coded for privacy protection

REFERENCES:
- [Background] Basaran B, Basaran A, Kozanhan B, Kasdogan E, Eryilmaz MA, Ozmen S. Analgesia and respiratory function after laparoscopic cholecystectomy in patients receiving ultrasound-guided bilateral oblique subcostal transversus abdominis plane block: a randomized double-blind study. Med Sci Monit. 2015 May 7;21:1304-12. doi: 10.12659/MSM.893593. PMID 25948166
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Ganapathy S, Sondekoppam RV, Terlecki M, Brookes J, Das Adhikary S, Subramanian L. Comparison of efficacy and safety of lateral-to-medial continuous transversus abdominis plane block with thoracic epidural analgesia in patients undergoing abdominal surgery: A randomised, open-label feasibility study. Eur J Anaesthesiol. 2015 Nov;32(11):797-804. doi: 10.1097/EJA.0000000000000345. PMID 26426576
- [Background] Lissauer J, Mancuso K, Merritt C, Prabhakar A, Kaye AD, Urman RD. Evolution of the transversus abdominis plane block and its role in postoperative analgesia. Best Pract Res Clin Anaesthesiol. 2014 Jun;28(2):117-26. doi: 10.1016/j.bpa.2014.04.001. Epub 2014 May 9. PMID 24993433